CLINICAL TRIAL: NCT04636294
Title: Follow-up of Patients With a Borderline COVID-19 PCR Test Result
Brief Title: Borderline COVID-19 PCR Test Result
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: f/2020/166
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Virus
MeSH Terms: conditions — COVID-19; Virus Diseases | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 suspected by symptoms, after high-risk contact or after a borderline PCR result.
  Interventions: Diagnostic Test: SARS-CoV-2 PCR

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 PCR — SARS-CoV-2 PCR of nasopharyngeal lysate.

SUMMARY:
Follow-up of patients with a borderline PCR result. Data of patients that were re-tested within 96 hours after receiving a borderline COVID-19 PCR result are reviewed.

This is a retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Every individual that delivers a nasopharyngeal lysate for SARS-CoV-2 RNA determination by PCR.

Exclusion Criteria:

* Patients without a previous borderline COVID-19 PCR result within 96 hours are excluded for the follow-up study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Ambulant (majority)
  * Hospital personnel
  * Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Ratio of positivity conversion after receiving a COVID-19 borderline PCR result. | 3 days

SECONDARY OUTCOMES:
Symptoms predicting COVID-19 positivity conversion after receiving a borderline PCR result. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Laboratory Jessa Hospital, Hasselt, Limburg, Belgium

REFERENCES:
- [Derived] Boeckmans J, Cartuyvels R, Hilkens P, Bruckers L, Magerman K, Waumans L, Raymaekers M. Follow-up testing of borderline SARS-CoV-2 patients by rRT-PCR allows early diagnosis of COVID-19. Diagn Microbiol Infect Dis. 2021 Jun;100(2):115350. doi: 10.1016/j.diagmicrobio.2021.115350. Epub 2021 Feb 18. PMID 33689985